CLINICAL TRIAL: NCT00781053
Title: Open Label Extension (OLE) for the Patients Treated in the ISD002-P144-07 Study With P144 Topical Adminsitration for Skin Fibrosis in Patients With Systemic Sclerosis
Brief Title: Open Label Extension (OLE) for the Patients Treated in the ISD002-P144-07 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ISDIN (Industry)
Collaborators: Digna Biotech S.L. (Industry)
Responsible Party: ISDIN, ISDIN
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISD003-P144-08; 2008-001265-28
Record Dates: First submitted 2008-10-24; First posted 2008-10-28 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Skin Fibrosis
Keywords: skin fibrosis; systemic scleroderma; systemic sclerosis; p144; orphan drug
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P144 cream (Experimental): P144 cream 0.03% will be used once a day during the whole extension period of 6 months.
  Interventions: Drug: P144 cream

INTERVENTIONS:
Drug: P144 cream — P144 cream 0.03% will be used once a day during the whole extension period of 6 months. The patient will apply the cream by him/herself or with a help of a person uniformly in a 10% maximum affected surface until absorption

SUMMARY:
Transforming growth factor-beta 1 is consistently over expressed in most fibrotic diseases and displays a variety of profibrotic effects in fibroblasts(25, 26). Activation of TGF-beta receptors induces the activation of several kinase signalling cascades leading to the phosphorylation of SMAD proteins as well as to the activation of SMAD-independent kinases that collectively activate ECM synthesis and fibroblast growth and differentiation into myofibroblasts. TGF-beta 1 i one of the main mediators in the fibrotic process, associated to both scarring and a long list of pathologies related to chronic inflammation and which affect all type of organs and tissues. An increase in TGF-beta1 mRNA and protein levels has been described in these processes. Peptide 144 (P144)is a acetic salt of a 14mer peptide from human TGF-beta1 type III receptor (betaglycan). P144 TGF-beta1-inhibitor has been specifically designed to block the interaction between TGF-beta1 and TGF-beta1 type III receptor, thus blocking its biological effects. P144 has shown significant antifibrotic activity in mice receiving repeated sucutaneous injections of bleomycin, a widely accepted animal model of human scleroderma, and could contribute to the development. The aim of the study is to asses the long-term safety of topical application of P144 cream in the treatment of skin fibrosis in patients with systemic sclerosis in an extension open-label treatment period of 6 additional months.

DETAILED DESCRIPTION:
Systemic sclerosis or scleroderma is a multisystemic disorder characterized by the excessive synthesis and deposition of extracellular matrix proteins that result in the fibrosis of skin and visceral organs (including gastrointestinal tract, lungs, heart and kidneys).The pathogenesis of scleroderma is complex and still poorly understood, but major pathways involved in the development of the condition are microvascular and immunological abnormalities, as well as dysregulation of fibroblast activity. One of the key molecules involved in the pathogenesis of skin fibrosis is the TGF-beta1; TGF-beta1 is a cytokine directly responsible for fibroblasts proliferation and collagen and extracellular matrix overproduction. The affected skin of patients with systemic sclerosis gradually becomes firm, thickened and eventually tightly bound to underlying subcutaneous tissue (indurative phase). It loses hair, oil, and sweat glands becoming dry and coarse. Changes begin distally in the extremities and advance proximally. Lesions develop over a period of time varying from months to a few years. In patients with limited scleroderma, only the skin of fingers, hands, face and lower arms and legs are affected. On the contrary, patients with the diffuse cutaneous disease, skin changes will become generalized, involving initially the extremities and followed by the face and trunk. Rapid progression of these changes over a 2 to 3 year period is usually associated with a greater risk of visceral disease. After several years of disease, the skin may soften and return to normal thickness or become thin and atrophic. The EMEA and FDA have granted P144 the orphan drug status for the treatment of systemic sclerosis. The primary objective is to assess the long-term safety of P144 crem topically administered in skin manifestations of systemic sclerosis patients in terms of the incidence of treatment related adverse events during the extension period of six months.

ELIGIBILITY:
Inclusion Criteria:

1. Previous participation and finalization of treatment period of the ISD002-P144-07 study without clinical relevant safety issues medically evaluated by the investigator.
2. For female subjects with childbearing potential: use of a known highly effective method of birth control, defined as those which results in a low failure rate: i.e. less 1% per year, (contraceptive pills, intrauterine contraceptive device, implants, vasectomized partner or sexual abstinence), for at least the extension study period and one month after the end of the extension study.
3. For male subjects with partners of childbearing potential:

   use of appropriate contraceptive methods (vasectomy, condoms or sexual abstinence), for at least the extension study period and one month after the end of the extension study.
4. Stable therapy for at least one month, except in the case of patients under treatment with putative disease modifying agents (immunosupressants like cyclophosphamide, or azathioprine) that will need at least three months of stable therapy, without the expectation of treatment modifications during the trial period..
5. Capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol specific procedures are performed

Exclusion Criteria:

1. Other skin diseases affecting the treatment area which could have been diagnosed during the ISD002-P144-07 study.
2. Woman became pregnant during the ISD002-P144-07 study.
3. Any new diagnosis since the ISD002-P144-07 study which includes: systemic sclerosis sine scleroderma, localized escleroderma, eosinophilic fascitis, or eosinophilia myalgia syndrome; any other definable connective tissue disease, such as rheumatoid arthritis, systemic lupus erythematosus, polymyositis, or dermatomyositis; clinically significant overlap condition; significant existing internal organ damage as defined in the guidelines for clinical trials in systemic sclerosis; history of skin cancer; other skin diseases affecting the treatment area.
4. Substantial history of environmental exposure to tainted rapeseed oil, vinyl chloride, L- tryptophan, bleomycin, trichoroethylene, or silica; PUVA therapy within 1 month of study drug initiation; concurrent interventional therapy that might independently influence outcome of trial, such as D-penicillamine, cyclosporine, methotrexate, interferon-γ or photopheresis; topical corticosteroids treatment affecting the selected area; cosmetics over the treatment area.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Assess the long-term safety of digna P144 cream topically administered in skin manifestations of systemic sclerosis patients. | 6 months

SECONDARY OUTCOMES:
Quality o life assessment, skin induration and hardness. In a subgroup of patients pharmacokinetic and elasticity will be measured. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Matucci, MD, PhD, Study Chair — University of Florence
Locations (17):
- Germany (4):
  - Herz- und Rheumazentrum Kerckhoff-Klinik, Bad Hauheim, Bad Hauheim
  - Klinikum der Johan Wolfgang Goethe-Universitat, Frankfurt, Frankfurt
  - Klinik und Poliklinik für Dermatologie und Vererologie, Cologne, Köln
  - Allergie-Centrum-Charité, Abteilung für, Berlin, State of Berlin
- Immunologiai es Reumatologiai Klinika, Pécs, Pécs, Hungary
- Azienda Ospedaliera Universitaria Careggi, Florence, Italy
- Poland (5):
  - Centrum Mirada, Bialystok, Bialystok
  - Samodzielny Publiczny Szpital Kliniczny, Katowice, Katowice
  - Katedra i Klinika Raumatologizno, Poznan, Poznan
  - Gabinet Lekarski Internistyczno- Reumatologiezny, Wroclaw, Wroclaw
  - Klinika Ftizjopneumonologii SAM, Zabrze, Zabrze
- Spain (3):
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid, Madrid
  - Clinica de Navarra, Pamplona, Pamplona
- United Kingdom (3):
  - Chapel Allerton Hospital, Leeds, Leeds
  - Royal Free Hospital, London, London
  - University Hospital Aintree, Liverpool

REFERENCES:
- See also: ISDIN exists to take care of the skin with reliable and scientifically tested products. — http://www.isdin.com